CLINICAL TRIAL: NCT03528733
Title: Feasibility of Single Exposure Dual Energy Subtraction With a Multi-Energy Digital Radiography Detector for Lung Lesions Detection
Brief Title: Feasibility of Multi-Energy Digital Radiography Detector for Lung Lesions Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KA Imaging Inc. (Industry)
Collaborators: Grand River Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KAIGRH1
Record Dates: First submitted 2018-05-04; First posted 2018-05-18 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Lung Tumor; Solitary Pulmonary Nodule
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-Energy Detector (Experimental): Multi-Energy Digital Radiography Detector System
  Interventions: Device: Multi-Energy Digital Radiography Detector System

INTERVENTIONS:
Device: Multi-Energy Digital Radiography Detector System — A Multi-energy digital flat panel detector for Single Exposure Dual-Energy Subtraction radiography is developed to capture x-ray images with improved tissue differentiation. Tissue-selective images can be produced at various tissue levels such as bone and soft tissue to visualize obscured anomalies that are not apparent to General Radiography.
  Other Names: Multi-Energy X-ray Detector

SUMMARY:
A single-centre, industry sponsored, pilot study to assess the feasibility of Single Exposure Dual Energy Subtraction with a Multi-Energy digital radiography detector as an imaging platform for lung lesion detection.

DETAILED DESCRIPTION:
A feasibility study is proposed to investigate the imaging characteristics captured by a Single Exposure Dual-Energy Subtraction digital radiography with KA Imaging's Multi-energy detector.

The acquisition of Dual-Energy Subtraction radiography will consist of using the Multi-Energy detector integrated into the X-ray system in Grand River Hospital. Patient will receive a Multi-Energy Chest radiography exam on the same day as their routine chest CT exam. Each Multi-Energy radiography exam will consist of one Chest PA image and one Chest LAT image. Duration of each procedure is 60 minutes. The Multi-Energy Detector will generate a General Radiography Image and Dual-Energy Subtracted Images.

Visualization of lung lesions by Multi-Energy detector will be compared to corresponding CT exam and general radiography results. Imaging data will be evaluated qualitatively by radiologists on data collection form to describe the findings on the images. Further comparison between general radiography, Dual-Energy Subtraction radiography and CT will be analyzed to determine the differences of imaging characteristics such as description of image quality and visibility of relevant anatomical structures and anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Patients with previously diagnosed carcinoma with lung metastases, or patients with previously detected lung nodule
* Subject is able to provide informed consent
* Study participant is scheduled to have a chest CT exam as part of their routine care.
* Study participant is able to stand and be still during the exams.

Exclusion Criteria:

* Not able or willing to provide Informed Consent, or consent is withdrawn.
* Study participant is pregnant
* Study participant is unable to perform standard radiography exam and CT exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Multi-Energy images will be compared to baseline Chest CT images for visualizing lung lesions. | 3 months
  Multi-Energy images will be compared to baseline Chest CT images for visualizing lung lesions, as determined. Expert readers will qualitatively evaluate the imaging differences (e.g. motion artifacts, technical defects, ease of anomalies identification, etc) with an evaluation form with a questionnaire grading system (i.e. 1 (severe defect), 2 (moderate defect) to 5 (no defect)).

SECONDARY OUTCOMES:
Multi-Energy images will be compared to standard radiography images for visualizing lung lesions. | 3 months
  Multi-Energy images will be compared to standard radiography images for visualizing lung lesions, as determined. Expert readers will qualitatively evaluate the imaging differences (e.g. motion artifacts, technical defects, ease of anomalies identification, etc) with an evaluation form with a questionnaire grading system (i.e. 1 (severe defect), 2 (moderate defect) to 5 (no defect)).

CONTACTS AND LOCATIONS:
Locations (1):
- Grand River Hospital, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No